CLINICAL TRIAL: NCT02062736
Title: Studio Osservazionale Per Valutare l'Adeguatezza Del Dosaggio Del Metadone, Nelle Terapie di Mantenimento, in Rapporto Agli Obbiettivi di Outcome, in Pazienti Tossicodipendenti da Eroina. (METODO)
Brief Title: Observational Study to Assess the Adequacy of Methadone Dosage, in Heroin Addicted Patients in a MMT.
Acronym: METODO
Status: Completed | Type: Observational
Sponsor: L.Molteni & C. dei F.lli Alitti-Soc. di Esercizio S.p.A. (Industry)
Collaborators: Solaris CRO (Industry)
Responsible Party: Sponsor
Other Study IDs: M.E.T.O.D.O.
Record Dates: First submitted 2014-01-24; First posted 2014-02-14 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Heroin Addiction
Keywords: methadone; heroin addiction; methadone maintenance treatment; adequate dosage of methadone
MeSH Terms: conditions — Heroin Dependence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pts addicted to heroin in MMT: patients addicted to heroin who have undertaken methadone maintenance treatment

SUMMARY:
The purpose of the study ( observational and prospective ) is to evaluate the efficacy and tolerability of the methadone maintenance treatment in patients addicted to heroin. The efficacy and tolerability are assessed by correlating to the adequacy of the dosage of methadone. The patients will be observed for two years.

DETAILED DESCRIPTION:
500 patients will be selected among all patients addicted to heroin according to DSM-IV_TR (Diagnostic and Statistical Manual of Mental Disorders IV_ text revision), in maintenance methadone treatment, observed in the involved sites. The investigators will use treatment schemes with methadon conform to clinical practice and according to SPC (Summary of Product Characteristics).

The enrollment will be competitive. Patients that meet incl/excl and that sign the informed consent, will be observed for 2 years. Follow up visits will be performed according to routine procedures, for patients that belong regularly to site at 3/6/9/12/18/24 months post V1. During the visits, patients will be assessed by validated and used as clinical practice questionnaires . For the evaluations of tolerability and safety the laboratory tests and electrocardiograms routinely performed will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Over 18 years of age
* Patients with a diagnosis of heroin addiction according to ICD-10 (International Classification of Diseases)
* Patients who have undertaken a methadone maintenance treatment
* Adhesion to observational study by signing informed consent.

Exclusion Criteria:

* Inability to follow the observation
* Diagnosis of decompensated psychotic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients addicted to heroin and who have undertaken a methadone maintenance treatment, observed in involved centres.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-02; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
the efficacy of the methadone maintenance treatment in addicted heroin patients, evaluating the correlation among efficacy and adequate dosage in comparison to not adequate dosage. | 2 years ( 7 visits for patient )

SECONDARY OUTCOMES:
QT prolongation risk in patients addicted to heroin who have undertaken MMT | 2 years ( evaluation at t0, t0 +6/12/18/24 months)
psychopathological status of observed patients in correlation with the adequate dosage in comparison to not adequate dosages | 2 years ( 7 visits for patient )
pharmacoeconomic condition correlated with the adequate dosage in comparison to not adequate dosage. | 2 years ( 7 visits for patient )

CONTACTS AND LOCATIONS:
Overall Officials: Donatella Mariani, Study Chair — Solaris CRO
Locations (5):
- Italy (5):
  - Dipartimento DSM, DP area Dipendenze Patologiche, UOSD Ser.T BO est, Bologna, BO
  - Dipartimento delle Dipendenze ASL MI 2, Milan, MI
  - Servizio dipendenze, AUSL, Pescara, PE
  - Dipartimento Dipendenze, ASL TO 2, Torino, TO
  - U.O.C. Ser.T ASL RMC, Distretto 11, Roma

REFERENCES:
- [Background] D'Egidio PF, Bignamini E, De Vivo E, Leonardi C, Pieri MC, Gonzalez-Saiz F, Lucchini A; METODO Study Team. METODO, a prospective observational study to assess the efficacy and tolerability of methadone in heroin-addicted patients undergoing a methadone maintenance treatment: preliminary results at baseline evaluation. Subst Use Misuse. 2013 Dec;48(14):1530-40. doi: 10.3109/10826084.2013.800886. Epub 2013 Jul 3. PMID 23822738